CLINICAL TRIAL: NCT05753488
Title: The Effect of Biomarkers of Inflammation on Graft Function
Brief Title: The Effect of Biomarkers of Inflammation on Graft Function in Kidney Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, Principal investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-23-3250
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Renal Transplant Failure and Rejection; Inflammation
MeSH Terms: conditions — Rejection, Psychology; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ınflammation
  Interventions: Diagnostic Test: graft function
- non inflammation
  Interventions: Diagnostic Test: graft function

INTERVENTIONS:
Diagnostic Test: graft function — renal transplantation

SUMMARY:
The aim of the study was to investigate the relationship of inflammation markers with postoperative graft function and mortality in patients undergoing kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent renal transplantation

Exclusion Criteria:

* patient refusal

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients underwent renal transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
RDW | baseline
  Red Cell Distribution Width
PNI | baseline
  prognostic nutrition index (PNI) calculated as 10 × serum albumin (g/dl) + 0.005 × total lymphocyte count (per mm3)
De Ritis | baseline
  De Ritis described the ratio between the serum levels of aspartate transaminase (AST) and alanine transaminase (ALT)
graft function | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided